CLINICAL TRIAL: NCT03913442
Title: A Phase IV, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study of the Effects of Colchicine on Pain and Inflammation in Subjects With Knee Osteoarthritis
Brief Title: Colchicine for the Treatment of Osteoarthritis of the Knee
Acronym: CLOAK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01796
Record Dates: First submitted 2019-04-02; First posted 2019-04-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo in capsule identical to study drug
  Interventions: Drug: Placebo oral capsule
- Colchicine (Experimental): 0.6 or 0.8 mg orally once daily.
  Because recent studies suggest that a dose of 0.6mg may be sufficient for chronic inflammatory suppression and may reduce the already low risk of toxicity of 0.8mg, for the remainder (second half) of the study the dosage will be switched from 0.8mg to a 0.6mg dose to allow comparison of the two doses.
  Interventions: Drug: Colchicine 0.8 mg or 0.6 mg orally once daily

INTERVENTIONS:
Drug: Colchicine 0.8 mg or 0.6 mg orally once daily — Colchicine 0.8 mg orally once daily for 1.5 months, and then 0.6 mg once daily for the remainder of the time (1.5 months)
  Arms: Colchicine
Drug: Placebo oral capsule — Placebo 0.8 mg or 0.6 mg orally once daily for 3 months
  Arms: Placebo

SUMMARY:
This prospective, double-blinded, placebo-controlled, randomized trial will enroll 120 SKOA subjects at the NYU Center for Musculoskeletal Care. Patients meeting entry criteria will be randomized 1:1 to treatment with colchicine or placebo daily for 3 months. Subjects will have detailed evaluation of standardized clinical pain outcomes, candidate peripheral blood biomarkers, baseline knee radiographs as well as MSK-US, and a subset will undergo evaluation of their synovial fluid.

ELIGIBILITY:
Inclusion Criteria:

* Are 40 years old or older
* Continue to experience frequent knee symptoms as defined above
* Have KL grade 2 or 3 on their last knee radiograph done for the parent study
* Have an estimated glomerular filtration rate (eGFR) > 30 ml/min (MDRD equation) and liver transaminases < 2x the upper limit of normal
* Have a BMI ≤ 32 at the time of enrollment
* Agree to be randomized to take colchicine or placebo daily for 3 months

Exclusion Criteria:

* Have received hyaluronic acid or corticosteroid steroid injection within the past 3 months
* Have a diagnosis of gout/pseudogout or other inflammatory arthritis (rheumatoid arthritis, psoriatic arthritis, reactive arthritis, spondyloarthropathy etc).
* Have a diagnosis of diabetes mellitus, chronic infectious disease, congestive heart failure, non-cutaneous cancer within the past 5 years
* Plan on undergoing total knee replacement within the next 3 months
* Be using any medication that is a strong CYP3A4 inhibitor whose metabolism may interact with colchicine (e.g., certain protease inhibitors, certain azole antifungal agents, clarithromycin).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Pillinger, MD, FACP, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Michael.pillinger@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Colchicine: 0.6 or 0.8 mg orally once daily.
  Because recent studies suggest that a dose of 0.6mg may be sufficient for chronic inflammatory suppression and may reduce the already low risk of toxicity of 0.8mg, for the remainder (second half) of the study the dosage will be switched from 0.8mg to a 0.6mg dose to allow comparison of the two doses.
  Colchicine 0.8 mg or 0.6 mg orally once daily: Colchicine 0.8 mg orally once daily for 1.5 months, and then 0.6 mg once daily for the remainder of the time (1.5 months)
Period: Overall Study
Arm/Group | Placebo | Colchicine
Started | 60 | 60
Completed | 51 | 49
Not Completed | 9 | 11
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Terminations | 2 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Colchicine | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.3) | 66.1 (10) | 66.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 41 | 37 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 33 | 30 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Pain Score
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | -1.45 (2.45) | -1.16 (2.22)

2. Secondary Outcome: Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Score
Description: The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms/stiffness (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The KOOS Pain Score refers to a specific subscale within the KOOS questionnaire that measures the severity of knee pain experienced by a patient, consisting of nine questions where each response is scored on a scale from 0 (no pain) to 4 (extreme pain), with a higher score indicating greater pain intensity; the overall pain score is then calculated as a percentage of the maximum possible score, where 0 represents the worst possible pain and 100 represents no pain at all.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 9.5 (20) | 5.2 (19)

3. Secondary Outcome: Change in the KOOS Stiffness Score
Description: The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms/stiffness (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). Each item on the KOOS is scored on a scale from 0 (no problems) to 4 (extreme problems), and then the scores are calculated to generate a final score between 0 and 100. The KOOS stiffness score is a percentage from 0 to 100 that measures how much stiffness a patient experiences in their knee. A score of 0 indicates the most stiffness, while a score of 100 indicates no stiffness.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 6.6 (15.7) | 5.5 (19.1)

4. Secondary Outcome: Change in the KOOS Physical Function Score
Description: The KOOS's five patient-relevant dimensions are scored separately: Pain (9 items); Symptoms/Stiffness (7 items); Function, Daily Living (17 items); Function, Sports and Recreational Activities (5 items); Quality of Life (4 items). The KOOS Physical Function items are scored on a Likert scale from 0 to 4, with 0 indicating no problems and 4 indicating extreme problems. The scores for each dimension are then transformed to a scale from 0 to 100, where 0 represents extreme problems with knee function and 100 indicates no problems at all.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 9.8 (17.6) | 7.4 (17.5)

5. Secondary Outcome: Change in the KOOS Quality of Life Score
Description: The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms/stiffness (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). A KOOS Quality of Life score ranges from 0 to 100, where 0 represents the worst possible knee-related quality of life and 100 indicates no problems at all. A higher score indicates better quality of life related to the knee.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 6.9 (22) | 3.5 (15.8)

6. Secondary Outcome: Change in the KOOS Sports and Recreational Activities
Description: The KOOS's five patient-relevant dimensions are scored separately: Pain (9 items); Symptoms/Stiffness (7 items); Function, Daily Living (17 items); Function, Sports and Recreational Activities (5 items); Quality of Life (4 items). The KOOS Sports and Recreational Activities 9 items are scored on a Likert scale from 0 to 4, with 0 indicating no problems and 4 indicating extreme problems relating to sports and recreational activities. The scores are then transformed to a scale from 0 to 100, with 100 indicating no knee problems with sports and recreational activities and 0 indicating extreme knee problems with sports and recreational activities .
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 0.0 (25.8) | 2.8 (19.4)

7. Secondary Outcome: Change in the KOOS Total Score
Description: The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms/stiffness (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
score on a scale | 6.5 (20.7) | 4.9 (18.1)

8. Secondary Outcome: Number of Participants Who Used Acetaminophen or Other Medications for Pain
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
Participants | 15 | 13

9. Secondary Outcome: Number of Participants Who Used Acetaminophen or Other Medications for Pain
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
Participants | 16 | 12

10. Secondary Outcome: Change in Number of Participants Who Used Acetaminophen or Other Medications for Pain
Time Frame: 6 weeks, 3 months
Measure: Number; unit: participants
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
participants | -1 | 1

11. Secondary Outcome: Change in Inflammatory Plasma Marker: Interleukin-1 Receptor Antagonist (IL-1Ra)
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
pg/mL | -66 (231.9) | -7.3 (194)

12. Secondary Outcome: Change in Inflammatory Plasma Marker: Prostaglandin E2 (PGE2)
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
pg/mL | 100 (586.4) | 72.4 (737.3)

13. Secondary Outcome: Change in Musculoskeletal Ultrasound (MSK-US)-Measured Effusion
Description: Size of effusion is measured as millimeters
Time Frame: Baseline, 3 months
Population: In lieu of synovitis whose measurements proved difficult, the team relied on MSK-US-measured effusions. Only 28 and 19 participants effusion data were collected for the placebo and colchicine group, respectively.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 28 | 19
millimeter | -1.2 (2.4) | -1.5 (3.0)

14. Secondary Outcome: Change in Rates of Crystal Deposition (Urate, Calcium) on MSK-US
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
mg/dL | 0 (0) | 0 (0)

15. Secondary Outcome: Change in Inflammatory Plasma Marker: Highly Sensitive C-reactive Protein (hsCRP)
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
mg/L | 0.1 (4.1) | -4.7 (15.6)

16. Secondary Outcome: Change in Inflammatory Plasma Marker: Uric Acid
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Colchicine
Number analyzed (Participants) | 51 | 49
mg/dL | 0.2 (0.7) | -0.8 (1.0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Placebo | Colchicine
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 34/51 | 36/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Colchicine (N=49)
Loose stools (Gastrointestinal disorders) | 11 | 19
Abdominal discomfort (Gastrointestinal disorders) | 7 | 2
Nausea/ Vomiting (Gastrointestinal disorders) | 5 | 4
Headache (General disorders) | 6 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03913442/Prot_SAP_000.pdf